CLINICAL TRIAL: NCT02364778
Title: ORBID Trial: Three-Dimensional (3D) Optical Coherence Tomography Guided Assessment of Side Branch Vessel After Provisional Main Vessel Stenting in Coronary Artery Stenting
Brief Title: Single-centre, Registry Trial, the Patients Presented With Stable Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Annapoorna Kini, Professor, Medicine, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 14-1777
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Results first posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Artery Disease
Keywords: CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Provisional stenting strategy: Patients with stable coronary artery disease with angiographic main vessel lesion not involving side branch (SB) in whom provisional stenting strategy is planned.

SUMMARY:
This is a prospective study to analyze the outcome of provisional main vessel stenting on side branch by utilizing Two-Dimensional (2D) and Three-Dimensional (3D) frequency domain optical coherence tomography (FD-OCT). To analyze the fate of side-branch after provisional main vessel stenting based on morphology defined prior to PCI by OCT. Offline analysis of side branch impingement of the ostium of SB leading to acute loss in SB diameter area, carina shift and plaque shift will be also be performed.

DETAILED DESCRIPTION:
Patients with stable coronary artery disease with angiographic main vessel lesion not involving side branch (SB) in whom provisional stenting strategy is planned will be recruited. All the participants of the registry will receive same stent. OCT will be performed to analyze plaque morphology, SB size, SB angle and side branch ostial involvement.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age presenting with stable coronary artery disease.
* Angiographic lesion not involving side branch (SB) in whom provisional main vessel stenting strategy is planned after reviewing angiogram will be recruited

Exclusion Criteria:

* Patient with lesion involving side branch ( >70 %) by angiogram and need pre-dilation.
* Patients with ostial left main artery lesions or ostial right coronary artery lesions
* Female patients with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Known allergy to acetylsalicylic acid or clopidogrel.
* Planned surgery within 12 months.
* History of bleeding diathesis
* Major surgery within 15 days
* Life expectancy < 12 months.
* Patients with kidney dysfunction (CrCl<30)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable coronary artery disease with angiographic main vessel lesion not involving side branch (SB) in whom provisional stenting strategy is planned
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annapoorna Kini, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Kini AS, Vengrenyuk Y, Pena J, Yoshimura T, Panwar SR, Motoyama S, Kezbor S, Hasan CM, Palkhiwala S, Kovacic JC, Moreno P, Baber U, Mehran R, Narula J, Sharma SK. Plaque morphology predictors of side branch occlusion after provisional stenting in coronary bifurcation lesion: Results of optical coherence tomography bifurcation study (ORBID). Catheter Cardiovasc Interv. 2017 Feb 1;89(2):259-268. doi: 10.1002/ccd.26524. Epub 2016 Mar 31. PMID 27029714

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Provisional Stenting Strategy
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study group consisted of 30 patients with 30 bifurcation coronary lesions that did not involve SB ostium.
Groups:
- SB Ostium DS >50%: Side branch (SB) ostium diameter stenosis (DS) >50%
- SB Ostium DS ≤50%: Side branch (SB) ostium diameter stenosis (DS) ≤50%
- Total: Total of all reporting groups
Arm/Group | SB Ostium DS >50% | SB Ostium DS ≤50% | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (2.5) | 63.1 (2.2) | 63.6 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 7 | 14 | 21
Hypertension [Number; unit: participants]
  yes | 9 | 15 | 24
  no | 1 | 5 | 6
Dyslipidemia [Number; unit: participants]
  yes | 9 | 19 | 28
  no | 1 | 1 | 2
Diabetes mellitus [Number; unit: participants]
  yes | 5 | 8 | 13
  no | 5 | 12 | 17
Current smoking [Number; unit: participants]
  yes | 2 | 2 | 4
  no | 8 | 18 | 26
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (2.0) | 31.5 (2.2) | 30.3 (1.6)
Prior MI [Number; unit: participants] — Prior myocardial infarction history
  participants
    yes | 1 | 3 | 4
    no | 9 | 17 | 26
CCS angina grade III or IV [Number; unit: participants] — Canadian Cardiovascular Society (CCS)
  participants
    yes | 8 | 18 | 26
    no | 2 | 2 | 4
Statin use [Number; unit: participants]
  yes | 8 | 16 | 24
  no | 2 | 4 | 6
Antiplatelet therapy [Number; unit: participants]
  Clopidogrel | 5 | 17 | 22
  Prasugrel | 3 | 1 | 4
  Ticagrelor | 2 | 2 | 4
Total cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 136 [127 to 167] | 136 [127 to 168] | 136 [127 to 179]
HDL cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 41 [36 to 42] | 40 [32 to 52] | 41 [32 to 52]
LDL cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 72 [59 to 86] | 73 [58 to 92] | 72 [57 to 92]
Triglyceride [Median (Inter-Quartile Range); unit: mg/dL] | 107 [85 to 152] | 84 [61 to 151] | 102 [63 to 151]

OUTCOME MEASURES:

1. Primary Outcome: MLD SB Diameter
Description: Optical coherence tomography (OCT) - a high resolution intravascular imaging technique to assess side branch size. Side branch diameter will be measured by QAngio OCT software from Medis. Three-Dimensional Quantitative Coronary Angiography (3D-QCA) Analysis of Bifurcation Lesions Before (PRE) and After (POST) Provisional Stenting. Main vessel minimal lumen diameter (MLD)
Time Frame: day 1
Measure: Mean (Standard Error); unit: mm
Arm/Group | SB Ostium DS >50% | SB Ostium DS ≤50%
Number analyzed (Participants) | 10 | 20
mm
  PRE | 08. (0.1) | 1.0 (0.1)
  POST | 2.3 (0.1) | 2.2 (0.1)

2. Secondary Outcome: SB Angle
Description: Optical coherence tomography - a high resolution intravascular imaging technique to assess side branch (SB) angle. Side branch angle will be measured by QAngio XA 3D software (Medis). Three-Dimensional Quantitative Coronary Angiography (3D-QCA) Analysis of Bifurcation Lesions Before (PRE) and After (POST) Provisional Stenting. Bifurcation angles (BA)
Time Frame: day 1
Measure: Mean (Standard Error); unit: degree
Arm/Group | SB Ostium DS >50% | SB Ostium DS ≤50%
Number analyzed (Participants) | 10 | 20
degree
  PRE Proximal BA | 140.3 (6.0) | 147.7 (4.0)
  POST Proximal BA | 140.5 (7.2) | 141.5 (3.7)
  PRE Distal BA | 48.0 (3.6) | 49.9 (2.8)
  Post Distal BA | 47.9 (4.8) | 48.3 (2.6)

3. Secondary Outcome: SB Ostial Involvement
Description: Optical coherence tomography - a high resolution intravascular imaging technique to assess side branch ostial involvement. Side branch area will be measured by QAngio OCT software (Medis). Three-Dimensional Quantitative Coronary Angiography (3D-QCA) Analysis of Bifurcation Lesions Before (PRE) and After (POST) Provisional Stenting. Minimal lumen diameter (MLD)
Time Frame: day 1
Measure: Mean (Standard Error); unit: mm
Arm/Group | SB Ostium DS >50% | SB Ostium DS ≤50%
Number analyzed (Participants) | 10 | 20
mm
  PRE side branch ostium MLD | 1.4 (0.3) | 1.6 (0.1)
  POST side branch ostium MLD | 0.8 (0.1) | 1.8 (0.1)

4. Secondary Outcome: Diameter Stenosis (DS)
Description: Three-Dimensional Quantitative Coronary Angiography (3D-QCA) Analysis of Bifurcation Lesions Before (PRE) and After (POST) Provisional Stenting. Side Branch Ostium Diameter Stenosis (DS).
Time Frame: day 1
Measure: Mean (Standard Error); unit: percentage of 100
Arm/Group | SB Ostium DS >50% | SB Ostium DS ≤50%
Number analyzed (Participants) | 10 | 20
percentage of 100
  PRE DS | 30.0 (4.1) | 24.0 (3.2)
  POST DS | 63.1 (2.6) | 27.7 (3.5)

ADVERSE EVENTS:
Description: Adverse events information not collected
Arm/Group | SB Ostium DS >50% | SB Ostium DS ≤50%
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Small number of cases. Results represent a hypothesis-generating pilot study rather than a definitive result.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes